CLINICAL TRIAL: NCT00042679
Title: A Phase 2 Trial of Antisense Nucleotide to PKC-Alpha (LY900003, ISIS 3521) Plus Gemcitabine and Carboplatin in Patients With Advanced, Previously Untreated Non-Small Cell Lung Cancer.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 6429; H7X-MC-JVAB
Record Dates: First submitted 2002-08-02; First posted 2002-08-06 (Estimated); Last update posted 2006-07-19 (Estimated); Status verified 2006-07

CONDITIONS: Carcinoma, Non-Small-Cell Lung; Pulmonary Neoplasms; Neoplasms, Lung
Keywords: Non-Small-Cell Lung Cancer; Adenocarcinoma; Carcinoma Squamous; Adult Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms; Adenocarcinoma; Carcinoma, Squamous Cell | interventions — Gemcitabine; Carboplatin; ISIS 3521

INTERVENTIONS:
Drug: Gemcitabine
Drug: Carboplatin
Drug: LY900003

SUMMARY:
The purposes of this study are to determine the following:

Whether LY900003 plus gemcitabine and carboplatin can make your tumor smaller or disappear, and for how long.

If treatment with LY900003 plus gemcitabine and carboplatin can help you live longer.

The safety of LY900003 plus gemcitabine and carboplatin and any side effects that might be associated with the combination of these three drugs.

How LY900003 is distributed and broken down by your body when it is given with carboplatin and gemcitabine.

Whether LY900003 affects the way gemcitabine and carboplatin are distributed and broken down by your body.

DETAILED DESCRIPTION:
Definition: The phase 2 study will provide important information regarding effects of LY900003 on safety and efficacy of patients treated with gemcitabine and carboplatin. LY900003 will be given at approximately 2 mg/kg/day for the first 14 days of a 21-day cycle. The dose and schedule for LY900003 administration are based on results of prior studies of LY900003 and are currently being used in other studies of LY900003. Gemcitabine will be administered on Days 1 and 8 at 1250 mg/m2 and carboplatin will be given on Day 1 at AUC 5.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Non-Small-Cell Lung Cancer.
* Stage IV or Stage IIIB disease.
* ECOG Performance Status of 0 or 1.
* Adequate organ function
* One unidimensionally measurable lesion.

Exclusion Criteria:

* Prior therapy for NSCLC.
* Serious concomitant disorders.
* Untreated CNS metastases.
* Uncontrolled, active infection.
* Previous LY900003/ISIS trial participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2002-06

CONTACTS AND LOCATIONS:
Locations (11):
- United States (11):
  - Bakersfield, California
  - Berkeley, California
  - Torrance, California
  - Miami Beach, Florida
  - Chicago, Illinois
  - Park Ridge, Illinois
  - Baltimore, Maryland
  - Chattanooga, Tennessee
  - Lubbock, Texas
  - Charlottesville, Virginia
  - Milwaukee, Wisconsin